CLINICAL TRIAL: NCT03441568
Title: In-home Use Test of the New Modified Diprobase® Formulation to Assess the Safety and Tolerability in Infants and Children Under Physician's Control
Brief Title: In-home Use Test of the New Modified Diprobase Formulation to Assess the Safety and Tolerability in Infants and Children Under Physician's Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19690; 2017-004334-29 (EudraCT Number)
Record Dates: First submitted 2018-02-16; First posted 2018-02-22 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BAY987534 (Experimental): Infants and children with quiescent atopic dermatitis
  Interventions: Device: Modified Diprobase formulation (BAY987534)

INTERVENTIONS:
Device: Modified Diprobase formulation (BAY987534) — The modified Diprobase formulation will be applied topically twice daily over 14 days on the whole body and face.

SUMMARY:
To investigate the safety and tolerability of the modified Diprobase formulation over 14 days in infants and children with a history of Atopic Dermatitis (AD).

ELIGIBILITY:
* Children with normal or dry skin and a history of mild to moderate AD, but without any signs or symptoms within the last month prior to enrollment
* Skin type I - VI according to Fitzpatrick skin classification
* Aged 6 months to 48 months

Ages: 6 Months to 48 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2018-09-26 (Actual); Primary Completion 2019-08-02 (Actual); Study Completion 2019-08-02 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse event (AE) | Up to 14 days
Severity of adverse event | Up to 14 days
  The intensity of an AE is classified according to the following categories:
  * Mild
  * Moderate
  * Severe

CONTACTS AND LOCATIONS:
Locations (1):
- West Timperley Medical Centre, Altrincham, United Kingdom